CLINICAL TRIAL: NCT04582994
Title: The Role of Beta Oscillation in Mental Time Travel: a tACS Study in Healthy Subjects
Brief Title: The Role of Beta Oscillation in Mental Time Travel
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Goldsmiths, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: EC 1199
Record Dates: First submitted 2020-10-04; First posted 2020-10-12 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2021-04

CONDITIONS: Healthy Population
Keywords: Time Perception; Mental Time Travel; tACS; Brain Stimulation
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young participants: 30 young participants will perform the Mental Time Travel task while tACS stimulation is delivered at three different frequencies on the posterior parietal cortex. Interventions are administered in three different sessions in a pseudo-randomized order as described below:
  1. Day 1. Beta tACS (22Hz)
  2. Day 2. Alpha tACS (10 Hz)
  3. Day 3. Sham tACS
  Interventions: Behavioral: Beta tACS; Behavioral: Alfa tACS; Behavioral: Sham
- Old participants: 30 old participants will perform the Mental Time Travel task while tACS stimulation is delivered at three different frequencies on the posterior parietal cortex. Interventions are administered in three different sessions in a pseudo-randomized order as described below:
  1. Day 1. Beta tACS (22Hz)
  2. Day 2. Alpha tACS (10 Hz)
  3. Day 3. Sham tACS
  Interventions: Behavioral: Beta tACS; Behavioral: Alfa tACS; Behavioral: Sham

INTERVENTIONS:
Behavioral: Beta tACS — participants perform the Mental Time Travel task (duration 20 minutes), while tACS stimulation is delivered at Beta frequencies (22 Hz)
Behavioral: Alfa tACS — participants perform the Mental Time Travel task (duration 20 minutes), while tACS stimulation is delivered at Alfa frequencies (10 Hz)
Behavioral: Sham — participants perform the Mental Time Travel task (duration 20 minutes), while Sham tACS stimulation is delivered

SUMMARY:
The project aims to study the neural basis of Mental Time Travel (MTT), i.e. the ability to travel back and forth in time. It has been proposed that the self-projection in time is similar to the self-projection in space, emphasizing the role of spatial navigation in MTT. Indeed, the posterior parietal cortex, a key region for visual imagery in space-related tasks, and the temporo-parietal junction, a key region for mental projection, are both recruited by self-projection in time and space. However, the specific neural computation of the two processes remains unclear. One way to address this is by investigating the brain oscillations that may modulate MTT. One plausible candidate for MTT processing are beta oscillations because of their role in the production and perception of short temporal intervals, as opposed to alpha oscillations which correlate with illusory changes in self location in space. Thus, the present project investigates the hypothesis that MTT may rely on posterior parietal cortex's beta oscillations to self-project in time. Moreover, cause previous studies showed a different performance in time processing between young and elderly health population, we want to investigate also if there is a difference between these two populations in the capacity to travel mentally in time.

DETAILED DESCRIPTION:
A characteristic of human conscious experience is the ability to mentally project oneself to a new time location, either in the past or in the future, i.e. the so-called Mental Time Travel (MTT). The aim of the present project is to study the neural basis of MTT.

It has been proposed that the self-projection in time is similar to the self-projection in space, emphasizing the role of spatial navigation in MTT. Indeed, the posterior parietal cortex, a key region for visual imagery in space-related tasks, and the temporo-parietal junction, a key region for mental projection, are both recruited by self-projection in time and space. However, the specific neural computation of the two processes remains unclear. One way to address this is by investigating the brain oscillations that may modulate MTT. One plausible candidate for MTT processing are beta oscillations because of their role in the production and perception of short temporal intervals, as opposed to alpha oscillations which correlate with illusory changes in self location in space. Thus, we hypothesize that the MTT may rely on posterior parietal cortex's beta oscillations to self-project in time. Moreover, because previous studies showed a different performance in time processing between young and elderly health population, we want to investigate also if there is a differences between these two populations in the MTT.

To assess the MTT we developed a new task in which participants see stimulus faces of different ages, one at a time. Each face is presented with a short phrase describing a particular life event, commonly happening in middle age. Participants perform a 2-alternative forced choice: in the 'Past Projection', they indicate if it is likely or unlikely that the stimulus person has lived the life event 10 years ago; in the 'Future projection' that the stimulus person will live the event 10 years in the future. We use transcranial alternating current stimulation (tACS) to test within subjects the role of target (Beta) and control oscillations (Alpha), in addition to a control non-stimulation condition (Sham). To rule out that tACS may simply affect age perception, participants are also asked to report the age of each stimulus face (Age Estimation task). Moreover, to investigate if there is any correlation between the MTT and the perception of short temporal interval, participants perform a time reproduction task before the brain stimulation and the MTT task. In the Time Reproduction task, a blue square is presented with a variable duration (encoding phase). Immediately after the encoding phase, a red square of the same size and position is presented. Subjects press a response button when they considered that the same of the previously studied time interval has elapsed.

A pilot study from 11 participants shows that beta-tACS corresponds to a shift in the psychometric curve towards a younger age in the 'Past condition', and towards an older age in the 'Future condition'. Thus, participants indicated a younger face as more likely to have lived an event 10 years ago and an older face as more likely to live an event 10 years in the future. This suggests that beta-tACS leads to an under-estimation of time relative to sham and alpha-tACS. Crucially, there were no significant differences in estimating the veridical ages of the stimulus faces. Thus, beta oscillation may modulate self-projection in time, since these data are consistent with an under-estimation of time.

If confirmed, results will allow us to specify that self-projection in time relies on the posterior parietal regions and beta oscillations. Moreover, if supported by our future experiments involving space processing, this result may also shed a new light on the distinction between self-projection in space, which is known to rely on alpha, and self-projection in time that relies on beta. Overall, these data may point to the fact that beta oscillations are critical for processing long durations, in addition to their well-known role in supporting short durations. This may be because beta oscillation may serve as a memory standard to which different durations are compared.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-30 for the first group and age between 60-80 for the second group

Exclusion Criteria:

* • generalized cognitive impairment (score lower than 24 at the Mini Mental State Examination)

  * psychiatric disorders
  * additional neurological disorders
  * abusive use of alcohol or illicit drugs
  * Personal or familiar history of epileptic fits

Ages: 20 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Two groups of healthy partcipants. Age between 20-30 for the first group and age between 60-80 for the second group
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Change in Mental Time Travel Task. | at day 1, day 2 and day 3
  Participants see 420 stimulus faces of different ages, one at a time. Each face is presented with a short phrase describing a particular life event, commonly happening in middle age. Participants perform a 2-alternative forced choice: in the 'Past Projection condition', they indicate if it is "likely" or "unlikely" that the stimulus person has lived the life event 10 years ago, in the 'Future projection condition' that the stimulus person will live the event 10 years in the future. A psychometric curve will be computed on the proportions of Likely responses, both in the "Future-projection" and in the "Past-projection" condition. We will assess the change in performance between Alpha , Beta and Sham tACS stimulation. Beta-Alpha and Sham tACS stimulation will be delivered in a randomized order in three different days.

SECONDARY OUTCOMES:
Time Reproduction Task | at day 1
  In the Time Reproduction task, a blue square is presented with a variable duration (encoding phase) around a standard interval of 2000 ms (1600, 1800, 2000, 2200 and 2400 ms). Immediately after the encoding phase, a red square of the same size and position was presented. Subjects had to press a response button when they considered that the same (reproduction task) of the previously studied time interval had elapsed.
Change in Age Estimation task | at day 1, day 2, day 3
  Faces stimuli are presented one at time. Participants are asked to guess the age of the persons depicted on the screen. This is a control task to rule out the possibility that Brain stimulation may simply affect age perception. Thus we will assess the change in performance between the different sessions of tACS stimulation (at day 1, 2 and 3)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for study and reaserch in Cognitive Neuroscience, Cesena, ITA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anelli F, Avanzi S, Arzy S, Mancuso M, Frassinetti F. Effects of spatial attention on mental time travel in patients with neglect. Cortex. 2018 Apr;101:192-205. doi: 10.1016/j.cortex.2018.01.012. Epub 2018 Feb 2. PMID 29482017
- [Background] Arzy S, Collette S, Ionta S, Fornari E, Blanke O. Subjective mental time: the functional architecture of projecting the self to past and future. Eur J Neurosci. 2009 Nov;30(10):2009-17. doi: 10.1111/j.1460-9568.2009.06974.x. Epub 2009 Nov 11. PMID 19912333
- [Background] Wiener M, Parikh A, Krakow A, Coslett HB. An Intrinsic Role of Beta Oscillations in Memory for Time Estimation. Sci Rep. 2018 May 22;8(1):7992. doi: 10.1038/s41598-018-26385-6. PMID 29789611
- [Background] Lenggenhager B, Halje P, Blanke O. Alpha band oscillations correlate with illusory self-location induced by virtual reality. Eur J Neurosci. 2011 May;33(10):1935-43. doi: 10.1111/j.1460-9568.2011.07647.x. Epub 2011 Mar 13. PMID 21395867
- [Result] D'Angelo M, Frassinetti F, Cappelletti M. The Role of Beta Oscillations in Mental Time Travel. Psychol Sci. 2023 Apr;34(4):490-500. doi: 10.1177/09567976221147259. Epub 2023 Feb 16. PMID 37067986
- See also: D'Angelo M, Frassinetti F, Cappelletti M. The Role of Beta Oscillations in Mental Time Travel. Psychol Sci. 2023 Apr;34(4):490-500. doi: 10.1177/09567976221147259. Epub 2023 Feb 16. — https://pubmed.ncbi.nlm.nih.gov/37067986/